CLINICAL TRIAL: NCT00574470
Title: Anti Cytokine Combination Therapy With Daclizumab and Infliximab for Treatment of Steroid Refractory Acute GVHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Magalhaes-Silverman, Margarida, Clinical Professor, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200511718
Record Dates: First submitted 2007-12-14; First posted 2007-12-17 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Graft vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Daclizumab; Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Treatment with daclizumab/infliximab
  Interventions: Drug: daclizumab, infliximab

INTERVENTIONS:
Drug: daclizumab, infliximab — Daclizumab 1 mg/kg IV days 1, 4, 8, 15 and 22. Infliximab 10 mg/kg IV days 1, 8, 15 and 22.

SUMMARY:
The purpose of this study is to see whether serious graft versus host disease which is not well controlled with steroid treatment can be controlled with therapy with both daclizumab and infliximab. We hypothesize that a combination of daclizumab and infliximab will more effectively treat graft versus host disease than therapy with a single drug. The study also looks at whether chronic graft versus host disease develops, and survival at 6 and 9 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of steroid refractory aGVHD defined as no response to methylprednisolone at 2 mg/kg for 1 week or disease progression after 72 hours of methylprednisolone at this dose. Potential subject will have had no decrease in any GVHD organ staging as follows:

  * Skin rash, if present, does not decrease by one stage. This is based on the percent of the body involved with rash, plus presence of bullae and desquamation.
  * Gut GVHD, if present, does not decrease by one stage. This is based on volume of diarrhea, pain, and ileus.
  * Upper gastrointestinal GVHD, if present, does not resolve.
  * Liver GVHD, if present, does not decrease by one stage. This is based on total bilirubin level.
* Prior allogeneic hematopoietic stem cell transplantation using bone marrow, peripheral blood or umbilical cord cells. Recipients of standard as well as nonmyeloablative transplants are eligible.
* No previous immune suppressive therapy given for treatment of acute GVHD except for corticosteroids.
* Absolute neutrophil count greater than 0.5x106/L.
* Estimated creatinine clearance greater than 30 mL/minute.
* Written informed consent

Exclusion Criteria:

* Patient receiving either infliximab or daclizumab within seven days of study.
* Patient with uncontrolled infections will be excluded.
* Patients receiving other investigational agents for GVHD prophylaxis or treatment.
* Patients with congestive heart failure.
* Patients with history of intolerance/ hypersensitivity to daclizumab or infliximab.
* Age less than 18 years.
* Patients who are pregnant or at risk of pregnancy and unwilling to use acceptable birth control methods.
* Patients with an allergy to murine products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-01; Primary Completion 2007-11 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Complete or partial response of GVHD to treatment according to standard staging/grading scale | 28 days

SECONDARY OUTCOMES:
incidence of chronic GVHD and overall survival | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Margarida Silverman, MD, Principal Investigator — University of Iowa Hospitals
Locations (1):
- University of Iowa Hospitals, Iowa City, Iowa, United States